CLINICAL TRIAL: NCT02848118
Title: Capnography Monitoring the Hypoventilation During Bronchoscopic Sedation
Brief Title: Capnography Monitoring in the Bronchoscopic Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Lun Lo, MD, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 104-0872C
Record Dates: First submitted 2015-03-18; First posted 2016-07-28 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Hypoventilation
Keywords: Hypoventilation; capnography; bronchoscopy
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A nasal-oral cannula of capnography (Experimental): Start bronchoscopy when the nasal-oral capnography shows hypoventilation during bronchoscopic sedation.
  Interventions: Device: A nasal-oral cannula of capnography
- Sedation scale (Active Comparator): Start bronchoscopy when Observer Assessment of Alertness and Sedation scale (OAAS)=3~2 during bronchoscopic sedation.
  Interventions: Other: Observer Assessment of Alertness and Sedation scale

INTERVENTIONS:
Device: A nasal-oral cannula of capnography — After propofol infusion, the complete induction is defined when capnography shows hypoventilation and bronchoscope is then introduced to patients.
  Other Names: End-tidal CO2
  Arms: A nasal-oral cannula of capnography
Other: Observer Assessment of Alertness and Sedation scale — After propofol infusion, the complete induction is defined when OAAS is 3 to 2 (conscious sedation) and bronchoscope is then introduced to patients.
  Other Names: OAAS
  Arms: Sedation scale

SUMMARY:
Procedure sedation of flexible bronchoscopy (FB) comforts patients undergoing FB. Hypoventilation during FB is a concern. The investigators investigate the feasibility of monitoring capnography in FB sedation.

DETAILED DESCRIPTION:
Patients undergoing flexible bronchoscopy (FB) experience procedure-related symptoms. Current guidelines of FB recommend sedation to all patients undergoing FB, except when there are contraindications. Propofol or benzodiazepines plus an opioid are the common combination used to improve patient tolerance and satisfaction during FB. However, controversy about combining propofol and opioids persists because of the risk of over-sedation and cardiopulmonary depression.

While transition from alert into sedation during induction, like sleep, the respiratory drive and muscle tone of respiratory muscle and upper airway attenuate, which contribute hypoventilation and upper airway collapse, and further hypoxemia. Detection of cardiopulmonary depression traditionally has relied on continuous monitoring of heart rate, respiratory rate, and oxygen saturation. However, it has been shown that these monitors could not recognize hypoventilation early. Similar with other published data, around 40% of hypoxemia event occurred during FB sedation in our hospital. Further analysis of our data revealed around 15% event occurred during sedative induction.

Capnography is the noninvasive measurement of the partial pressure of carbon dioxide (CO2) from the airway during ventilation. The maximum partial pressure of CO2 obtained at the end of an exhaled breath is referred to as end-tidal CO2 (EtCO2). Studies have revealed the waveform analysis of capnography can provide early warning for prehypoxic respiratory depression in patients undergoing procedure sedation in emergency department and gastrointestinal endoscopy. Therefore, capnography can serve as a real-time measure of ventilatory status of sedative patients and the physicians could intervene before the occurrence of hypoxemia. Based on the advantage of non-invasive and real-time property of EtCO2 monitored by capnography, the investigators plan to conduct a clinical trial to evaluate if hypoxemia could be reduced by capnography of EtCO2 monitor during induction of FB sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective bronchoscopy and sedation

Exclusion Criteria:

* Age less than 18 years
* American Society of Anaesthesiologists (ASA) physical status classification IV or V
* Mallampati score of 4
* Severe sleep apnoea syndrome (apnoea-hypopnea index more than 40)
* Body mass index more than 42 in males or 35 in females
* Neurologic disorders or other conditions contributing to difficulty in assessing response
* Forced expiratory vital capacity (FVC) less than 15 ml/kg body weight, forced expiratory volume in one second (FEV1) less than 1000 ml, or FEV1/FVC less than 35%
* Chronic use of opioid drugs
* Pregnancy
* Patients with a known history of allergy to the study drugs, or to eggs, soybeans or sulfite products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | 60 minutes
  Oxyhemoglobin saturation less than 90% with any duration after induction to patient recovery.

SECONDARY OUTCOMES:
Patient satisfaction | 60 minutes
  A 10cm visual analogue scale about how the patients fell about the bronchoscopy
Patient cooperation accessed by bronchoscopists | 60 minutes
  A 10cm visual analogue scale about how the bronchoscopists fell the cooperation of patients during bronchoscopy.
Induction time | 10 minutes
  The length of time for achieving adequate sedative depth to start bronchoscopy
Procedure time | 30 minutes
  The length of time for complete bronchoscopy
Propofol dosage | 60 minutes
  the dose of propofol for induction and whole bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Lun Lo, MD, Principal Investigator — Chang Gung Medical fundation
Locations (1):
- Chung Gung Medical Fundation, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lin TY, Lo YL, Hsieh CH, Ni YL, Wang TY, Lin HC, Wang CH, Yu CT, Kuo HP. The potential regimen of target-controlled infusion of propofol in flexible bronchoscopy sedation: a randomized controlled trial. PLoS One. 2013 Apr 24;8(4):e62744. doi: 10.1371/journal.pone.0062744. Print 2013. PMID 23638141
- [Background] Soto RG, Fu ES, Vila H Jr, Miguel RV. Capnography accurately detects apnea during monitored anesthesia care. Anesth Analg. 2004 Aug;99(2):379-82, table of contents. doi: 10.1213/01.ANE.0000131964.67524.E7. PMID 15271710